CLINICAL TRIAL: NCT06346353
Title: Substance Consumption, Personality, and Cognitive Functioning of Chess Players and Non-chess Players - an Online Survey
Brief Title: Substance Consumption, Personality, and Cognitive Functioning of Chess Players
Status: Completed | Type: Observational
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Other Study IDs: Chess Cognition SUD
Record Dates: First submitted 2023-02-02; First posted 2024-04-04 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Addiction; Alcohol; Nicotine; Drugs; Personality; Depression; Anxiety
MeSH Terms: conditions — Behavior, Addictive; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chess players: Chess players who play tournament chess and have a DWZ (deutsche Wertungszahl) and/or ELO rating
- Non-chess players: Non-chess players or hobby chess players who do not have a DWZ or ELO rating

SUMMARY:
The aim of this project is to find out if there is a difference in addictive behavior, personality traits, and cognitive abilities between chess players and non-chess players.

DETAILED DESCRIPTION:
In the present planned study, tournament chess players will be compared with non-tournament chess playing individuals by means of an online survey. Among other things, the investigators want to investigate whether these groups of persons differ in various characteristics such as their consumption behavior (alcohol, tobacco, and drug use), their personality, their depressiveness and mood, or their cognitive abilities. The background is the question whether playing chess could be protective against substance use disorders or could mitigate the manifestation.

ELIGIBILITY:
Inclusion Criteria:

* all persons from the age of 18 years
* Inclusion in the group of chess players is based on the existence of a DWZ.
* Sufficient ability to answer the questionnaires

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The survey is aimed at people who are at least 18 years old. There is no upper age limit. There is a division into two groups. Firstly, people who play chess in a club and have a DWZ (German rating). Secondly, there is a comparison group of people who do not play chess or only play chess as a hobby and therefore do not have a DWZ.
Sampling Method: Non-Probability Sample
Enrollment: 756 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Substance Craving | baseline
  Mannheimer Craving Scale (MACS), Nakovics, Diehl, Geiselhart, & Mann, 2009
Alcohol Use | baseline
  Alcohol Use Disorders Indentification Scale (AUDIT-C), Bohn, Babor, & Kranzler, 1995
Automatic Alcohol Craving | baseline
  Craving Automated Scale - Alcohol (CAS-A), Vollstädt-Klein, Leménager, Jorde, Kiefer, & Nakovics, 2015
Severity of Nicotine Dependence | baseline
  Fagerstrom Test of Nicotine Dependence (FTND), Heatherton, Kozlowski, Frecker, & Fagerström, 1991
Automatic Cigarette Craving | baseline
  Craving Automated Scale - Cigarette Smoking (CAS-CS), Tan et al., 2022
Smoking Consequences | baseline
  Smoking Consequences Questionnaire (SCQ), Lewis-Esquerre, Rodrigue, & Kahler, 2005
Drug Abuse | baseline
  Drug Abuse Screening Test (DAST-10), Lam et al., 2015
Personality | baseline
  NEO five factor inventory (NEO-FFI), Körner et al., 2008
Depression | baseline
  Beck Depressions Inventar - II (BDI-II) Kühner, Bürger, Keller, & Hautzinger, 2007
Anxiety | baseline
  State Trait Anxiety Inventory (STAI - trait Version), Spielberger, 1983
self-efficacy | baseline
  Self-efficacy expectancy (SWE) Jerusalem & Schwarzer, 1999
coping with stress | baseline
  Brief COPE, Carver, Scheier, & Weintraub, 1989
Inhibition capacity | baseline
  Stop Signal Task (Sebastian et al., 2013)
Working Memory capacity | baseline
  N-back Task (Charlet et al., 2014)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Vollstädt-Klein, Prof. Dr., Principal Investigator — Central Institute of Mental Health, Mannheim
Locations (1):
- Klinik für Abhängiges Verhalten, Zentralinstitut für Seelische Gesundheit, Mannheim, Germany